CLINICAL TRIAL: NCT00328939
Title: Randomized, Single Blind, Parallel Study to Compare the Safety and Efficacy of ARIXTRA to Enoxaparine in Patients Undergoing Elective Major Hip or Knee Replacement or a Revision of Components.
Brief Title: ARIXTRA Local Study For Registration In China.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ITI105316
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Thromboembolism; Knee Replacement; Hip Replacement
Keywords: ARIXTRA; prevention of DVT
MeSH Terms: conditions — Thromboembolism

INTERVENTIONS:
Drug: ARIXTRA infusion
Drug: Enoxaparine infusion
  Other Names: ARIXTRA infusion

SUMMARY:
This is a local registration study in China to compare the safety and efficacy of ARIXTRA to Enoxaparine in patients undergoing elective major hip or knee replacement or a revision of components.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing either an elective major hip or knee replacement or revision.
* Signed written informed consent. Men or women of non-child bearing potential(i.e., post menopausal or with hysterectomy of bilateral tubule ligation) or women of childbearing potential without any plan to have a child.

Exclusion criteria:

* History of serious active bleeding in last 3 month
* Concurrent or history of thrombocytopenia ( Platelet< 100x109/L)
* History of hypersensitivity reaction to heparin, Low molecular weight heparin or pork product
* Acute bacterial endocarditis
* Congenital or acquired bleeding disease in last 3 months
* Concurrent uncontrolled ulcer or gastrointestinal disease with blood vessel dysplasia
* Concurrent hemorrhagic cerebrovascular disease or surgical history in cerebral, spine or eye
* Conditions need to leave a tubule in intradural or extradural
* Contraindication to anticoagulant or condition required to take long term oral anticoagulant
* Abnormality in hepatic (>1.5x UNL), renal (Clcr < 30ml/min) or cardiac function, uncontrolled hypertension or tumor Concurrent disorder of blood vessel in lower limb
* Positive result in Human Chorionic Gonadotropin test Participated in any other investigational study on Deep Vein Thrombosis prevention in last 90 days.
* Concurrently to have hip and knee or double hip/knee replacement at the same time

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2004-05

PRIMARY OUTCOMES:
Occurrence of overall DVT (deep vein thrombosis) events confirmed by ultrasound result within day 5-11 post operation.

SECONDARY OUTCOMES:
Occurrence of DVT with symptom and non-fatal PE (pulmonary embolism). Occurrence of fatal PE.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- China (7):
  - GSK Investigational Site, Zhengzhou, Henan
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Qingdao, Shandong
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai